CLINICAL TRIAL: NCT03057379
Title: State Immunization Information Systems to Improve HPV Vaccination Rates
Brief Title: HPV IIS Reminder/Recall- New York State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16-002040
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Reminder Systems
Keywords: HPV vaccine; Immunization registry; Reminder recall

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four arms to receive 0,1,2,or 3 reminders for overdue HPV vaccine doses.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control arm (No Intervention): Usual source of care
- 1 R/R per Dose (Experimental): Sending up to one recall notice per dose of HPV vaccine needed
  Interventions: Other: Vaccine Reminder Recall
- 2 R/R per dose (Experimental): Sending up to two recall notice per dose of HPV vaccine needed
  Interventions: Other: Vaccine Reminder Recall
- 3 R/R per dose (Experimental): Sending up to three recall notice per dose of HPV vaccine needed
  Interventions: Other: Vaccine Reminder Recall

INTERVENTIONS:
Other: Vaccine Reminder Recall — The investigators will be sending recall notices via phone call to 11-17 year olds who are eligible but lacking HPV vaccine doses recorded in the New York State Immunization Information System (NYSIIS). The investigators will be testing the effectiveness and cost effectiveness of up to 3 notices per dose with usual care (no intervention)
  Arms: 1 R/R per Dose; 2 R/R per dose; 3 R/R per dose

SUMMARY:
The overarching goal of this study is to evaluate the effectiveness, cost-effectiveness and sustainability of utilizing statewide Immunization Information Systems (IIS) to conduct centralized reminder/recall (R/R) to improve Human Papiloma Virus (HPV) vaccination rates among adolescents ages 11-17.

DETAILED DESCRIPTION:
The overarching goal of this study is to evaluate the effectiveness, cost-effectiveness and sustainability of utilizing statewide Immunization Information Systems (IIS) to conduct centralized reminder/recall (R/R) to improve HPV vaccination rates among adolescents ages 11-17. The investigators will extend previous research on effectiveness of centralized R/R to a new population--adolescents due for HPV vaccine-- and test the use of centralized R/R as a cancer-prevention strategy. Investigators will assess the effect of centralized R/R in two states--one with and one without mandated reporting of vaccinations to IISs, and disseminate IIS R/R to other states. Investigators will implement, evaluate (using the RE-AIM framework 31-36), and disseminate a collaborative, IIS-based centralized HPV vaccine R/R model in which partnerships of public health systems and primary care practices in two states (NY, CO) collaborate to remind parents about HPV vaccination.

Specific Aims and hypotheses:

Aim #1: Adapt IIS messages and delivery systems (e.g., algorithms) previously developed for centralized R/R for other vaccines to fit HPV vaccine IIS R/R.

Aim #2: Assess the impact and cost-effectiveness of centralized IIS-based (IIS-C) autodialer (phone) R/R in increasing vaccine rates [initial dose (HPV#1) and a complete series (HPV#3)] among teens.

Conduct a pragmatic trial, to assess the impact and cost effectiveness of centralized IIS-based (IIS-C) autodialer (phone) R/R in increasing initiation and completion rates for the HPV vaccine series in adolescents ages 11-17 years. The investigators will use a within-practice design, randomizing patients within randomly selected primary care practices to IIS-C R/R (1, 2, or 3 reminders per dose) compared to usual care (0 reminders from this study). The investigators will apply the RE-AIM framework to evaluate the reach, effectiveness/cost effectiveness, adoption, and implementation of IIS-C R/R.

Hypothesis 2a: IIS-C R/R will result in higher HPV vaccination rates than usual care.

Hypothesis 2b: IIS-C R/R will result in higher HPV vaccination rates than usual care in key subgroups (males and females, younger and older teens, urban//rural teens).

Hypothesis 2c: IIS-C R/R will be more cost-effective (cost/vaccine received) than usual care.

Aim #3: Disseminate IIS-C R/R across NY and CO and pilot in four IISs: (a) Develop an IIS-C HPV R/R toolkit, (b) Use a technical advisory group, (c) Initiate IIS-C R/R in four other IISs [Yr. 4].

By the end of the study investigators will have a feasible, sustainable, cost-effective model for HPV vaccine reminders that can be used nationally to prevent cervical cancer and other HPV-related cancers.

ELIGIBILITY:
Inclusion Criteria:

* 11 through 17 years of age
* patient of a participating practice (practices randomly selected)
* is either due for an HPV dose at baseline, or
* has initiated but not yet completed the HPV series at baseline

Exclusion Criteria:

* has completed the HPV vaccination series

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30616 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Initiation of the HPV vaccine series (receipt and documentation of initial dose of vaccine series within immunization registry) | 5 months from initial recall notices for the first dose
  Did the adolescent initiate the HPV vaccine series? The investigators are allowing up to 5 months after the initial recall notice for the adolescent to make an appointment and receive their dose. After that time frame, the investigators will not attribute vaccination to the recall. Receipt will be documented by providers within the state immunization registry via electronic medical record (EMR) direct transfer or manual entry.
Completion of the HPV vaccine series (receipt and documentation of final dose of vaccine series within immunization registry) | 5 months from first reminder received for last dose
  Did those eligible to complete the HPV vaccine series within the time frame of the study do so? The investigators are allowing up to 5 months after the first recall notice of the last dose (could be dose 2 or dose 3, depending on the age at which they received their first dose) for adolescents to complete their vaccination series. After that time frame, the investigators will not attribute vaccination to the recall. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry.

SECONDARY OUTCOMES:
Differences between arms - initiation | 5 months
  Is 1, 2, or 3 reminders per arm most effective and cost effective for initiation. Only those who need an initial dose at baseline will be eligible for this outcome. We will compare the arms (receipt of zero, 1, 2 or 3 reminders) to see if there are any differences between the arms in terms of receipt of the 1st dose of HPV vaccine
Differences between arms - completion | 20 months
  Is 1, 2, or 3 reminders per arm most effective and cost effective for completion. Because the second or third dose of the series is dependent on when the adolescent receives their initial dose, the investigators will be following eligible adolescents for 20 months to allow time for those who did not respond to the recall for the initial dose right away to be able to complete the series within the time frame. However, receipt of the completion dose will only be attributed to the recall if it was received within 5 months of the 1st recall for the completion dose. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California LA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided